CLINICAL TRIAL: NCT00882284
Title: Hydrocortisone Treatment of Hypotension in Term and Late Preterm Infants: An Observational Study
Brief Title: Hypotension in Neonates
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD-NRN-0040; U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD034216 (NIH); U10HD040492 (NIH); U10HD040689 (NIH); U10HD053089 (NIH); U10HD053109 (NIH); U10HD053119 (NIH); U10HD053124 (NIH); UL1RR024139 (NIH); UL1RR025744 (NIH); M01RR008084 (NIH)
Record Dates: First submitted 2009-04-01; First posted 2009-04-16 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Infant, Newborn; Hypotension; Blood Pressure
Keywords: NICHD Neonatal Research Network; Blood Pressure Management
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study collects information on the current incidence and management of hypotension in babies born at term or late preterm that are admitted to Neonatal Intensive Care Units (NICUs) within the Neonatal Research Network (NRN). Participants include all newborn infants born at 34 0/7 weeks gestation or greater who are admitted to NICU Network centers and intubated and mechanically ventilated at less than 72 hours of age. The information gathered will provide a framework for the design of a potential randomized controlled trial for the treatment of hypotension in neonates. This observational study is for a time-limited enrollment period of 4-6 months; NRN centers will continue to enroll until at least 50 patients are enrolled per center (for approximately 800-1,000 subjects total).

DETAILED DESCRIPTION:
An estimated 30-50 percent of infants born at or near term who require ventilation for respiratory failure also receive therapy for hypotension and associated clinical instability, such as poor urine output, poor circulation to the tissues, and metabolic acidosis (a pH imbalance in which the body accumulates too much acid). Emerging evidence, although limited, suggests that the underlying cause of hypotension in many of these infants is that their adrenal glands do not produce adequate amounts of cortisol.

This observational study is to determine the current incidence and management of hypotension in infants born at least 34 0/7 weeks gestation who are intubated and mechanically ventilated at less than 72 hours of age. The goal is to define a target population for a potential randomized controlled trial for the treatment of hypotension in such infants.

In this study, 16 NICHD Neonatal Research Network centers are enrolling at least 50 infants each, collecting basic demographic and baseline data on the mother and baby. In those infants treated for hypotension, data is collected on the dose, duration, and type of therapy, age and blood pressure at the time therapy is started, and the indication for the therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥34 0/7 weeks gestational age
* Intubated and mechanically ventilated within 72 hours of postnatal age

Exclusion Criteria:

* major congenital heart disease
* acute hypotension resulting directly from known acute maternal and/or fetal hemorrhage within 24 hours prior to delivery
* pituitary hypoplasia
* congenital adrenal hyperplasia
* known chromosomal disorders

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All newborn infants born at ≥34 0/7 weeks gestational age admitted to NICU Network centers who are intubated and mechanically ventilated within 72 hours of postnatal age
Sampling Method: Non-Probability Sample
Enrollment: 820 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of Hypotension in infants | < 72 hours of age until hospital discharge

SECONDARY OUTCOMES:
Management of hypotension in infants | < 72 hours of age through resolution of hypotension
Short-term outcomes, including: vasopressor/inotrope exposure, death, time to full nipple feedings, duration of ventilation, and length of NICU stay | < 72 hours of age until hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N Goldberg, MD, Principal Investigator — Duke University; Barbara J Stoll, MD, Principal Investigator — Emory University; Brenda B Poindexter, MD MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P Van Meurs, MD, Principal Investigator — Stanford University; Ivan D Frantz III, MD, Principal Investigator — Tufts Medical Center; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F Bell, MD, Principal Investigator — University of Iowa; Kristi L Watterberg, MD, Principal Investigator — University of New Mexico; Pablo J Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Roger G Faix, MD, Principal Investigator — University of Utah; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A Ehrenkranz, MD, Principal Investigator — Yale University
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/